CLINICAL TRIAL: NCT01408160
Title: A Phase 1 Study of the Deglycosylated Ricin A Chain-containing Combined Anti-CD19 and Anti-CD22 Immunotoxin Combotox in Combination With High-Dose Cytarabine in Adult Relapsed or Refractory B-lineage Acute Lymphoblastic Leukemia
Brief Title: Immunotoxin Therapy and Cytarabine in Treating Patients With Relapsed or Refractory B-Cell Acute Lymphoblastic Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Amit Verma, Principal Investigator, Albert Einstein College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-04-146; NCI-2013-01206 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 11-027; 11-04-146 (Other: Albert Einstein College of Medicine); P30CA013330 (NIH)
Record Dates: First submitted 2011-07-12; First posted 2011-08-03 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Adult B Acute Lymphoblastic Leukemia; Recurrent Adult Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Burkitt Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cytarabine; combotox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Combotox, cytarabine) (Experimental): Patients receive high-dose cytarabine IV over 2-3 hours every 12 hours on days 1-3 and deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins IV over 4 hours on days 8, 10, and 12. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Biological: Deglycosylated Ricin A Chain-Conjugated Anti-CD19/Anti-CD22 Immunotoxins; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Biological: Deglycosylated Ricin A Chain-Conjugated Anti-CD19/Anti-CD22 Immunotoxins — Given IV
  Other Names: Combotox
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I trial studies the side effects and the best dose of deglycosylated ricin A chain-conjugated anti-cluster of differentiation (CD)19/anti-CD22 immunotoxins when given together with cytarabine in treating patients with B-cell acute lymphoblastic leukemia that has come back after a period of improvement (relapsed) or does not respond to treatment (refractory). Immunotoxins, such as deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins, can find certain cancer cells and kill them without harming normal cells. Drugs used in chemotherapy, such as cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins with cytarabine may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) of Combotox (deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins) when added to high-dose cytarabine during salvage therapy for adult patients with relapsed or refractory B-lineage acute lymphoblastic leukemia.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of this regimen. II. To assess for the presence of a postulated CD34+/CD38-/low/CD19+ leukemic stem cell phenotype in the bone marrow at time of relapse and to assess its association with treatment outcome.

III. To determine the development of human mouse or ricin antibodies (human anti-mouse antibodies [HAMA]/human anti-ricin antibodies [HARA]).

IV. To determine the pharmacokinetic characteristics of Combotox. V. To evaluate the value of fractional excretion of sodium (FeNa) as early marker of toxicity.

OUTLINE: This is a dose-escalation study of deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins.

Patients receive high-dose cytarabine intravenously (IV) over 2-3 hours every 12 hours on days 1-3 and deglycosylated ricin A chain-conjugated anti-CD19/anti-CD22 immunotoxins IV over 4 hours on days 8, 10, and 12. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed B-lineage acute lymphoblastic leukemia (ALL) at diagnosis and either evidence of relapse/refractory disease based on a bone marrow/peripheral blood examination or evidence by cytogenetic studies or polymerase chain reaction (PCR) amplification; patients with only extramedullary disease in the absence of bone marrow or blood involvement are not eligible; patients with L3 (Burkitt's) are not eligible; for ALL in marrow or peripheral blood, immunophenotyping of the blood or marrow lymphoblasts must be performed to determine lineage (B cell, T-cell, or mixed B/T cell); NOTE: appropriate marker studies including CD19 (B cell), CD10, CD5, and CD7 (T cell) must be performed; co-expression of myeloid antigens (CD13 and CD33) will not exclude patients; if possible, the lineage specific markers cytoplasmic CD22 or CD79a (B cells), cytoplasmic CD3 (T cells) and cytoplasmic myeloperoxidase (MPO) (myeloid cells) must be determined; patients with mixed lineage ALL (ML-ALL) as defined by a lack of cytochemical markers of myeloid differentiation, and by the presence of immunophenotypic markers suggesting both lymphoid and myeloid differentiation, are allowed
* CD19 and/or CD22 must be expressed on at least 50% of the lymphoblasts
* Disease must be refractory to conventional induction therapy or relapsed after initial standard therapy for ALL; any number of prior therapies is permitted and including allogeneic and/or autologous stem cell transplant
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 2 months
* Total bilirubin =< 1.5 x institutional upper limit of normal, unless related to leukemic infiltration or hemolysis
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal, unless related to leukemic infiltration or hemolysis
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have recovered from effects of prior therapy; at least 2 weeks should have elapsed since the last dose of high dose chemotherapy; hydroxyurea, steroids and vincristine are allowed to control counts until eligibility is confirmed and study treatment can be initiated
* Adequate cardiac function defined as an ejection fraction of >= 50% by multi gated acquisition scan (MUGA) scan or echocardiogram and a corrected QT (QTc) interval of =< 450 ms for men and =< 460 ms for women
* Adequate pulmonary function defined as no evidence of dyspnea at rest
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 2 weeks (4 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Combotox or other agents used in study agents
* Presence of a significant pleural effusion by chest x-ray
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic
* Presence of active untreated central nervous system (CNS) leukemia
* Presence of graft-versus-host disease (GVHD) more than grade 2
* History of documented seizure disorder, presence of cerebellar dysfunction, dysphasia or altered mental status on neurological examination
* Human anti-mouse antibody (HAMA) levels of > 100 ug/ml or human ricin antibodies (HARA) > 100 ug/ml HARA after cycle 1
* Impaired liver function defined as a total bilirubin > 1.5 x normal range and AST or ALT > 2.5 x normal range unless secondary to Gilbert's disease, hemolysis or leukemic involvement of the liver
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with Combotox
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-06-26 (Actual); Study Completion 2018-06-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity, defined as grade 3 or greater non-hematological adverse event attributable to Combotox, graded per the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 28 days

SECONDARY OUTCOMES:
Clinical response rate (response defined as complete response or partial response) | Up to day 42
  Descriptive statistics and tabular representations will be used to describe and evaluate the response rates for each dose level.

OTHER OUTCOMES:
Change in expression of CD19 and CD22 on cell surface by flow cytometry | Baseline to up to day 42
  Evaluated as a percentage ranging from 0% to 100% of cells analyzed expressing the respective marker. The change in percentage expression from pre-treatment to post-treatment for cycle 1 only will be correlated with the response achieved. Response to treatment is defined as either complete or partial remission. The means of CD19 and/or 22 expression will be compared between the patients who showed response and those who didn't using a t-test if the data is normally distributed or otherwise the non-parametric alternative (Mann-Whitney U test).
Change in fractional excretion of urinary sodium (FeNa) | Day 0 to up to day 12
  Changes in the FeNa will be correlated to the development of grade 3 or greater vascular leak syndrome (VLS). VLS will be dichotomized into absent or mild (grade 0-2) versus moderate to severe (3-5). Changes in FeNa from baseline to day 8, 10 and 12 will be calculated as percent change at each time point. Associations will be tested for in a logistic regression model using presence of moderate or severe VLS as outcome as well as in a linear regression model using the grading of VLS as an ordinal variable. Both models will be adjusted for the use of diuretics and intravenous fluids.
Development of VLS | Up to day 12
  Changes in the FeNa will be correlated to the development of grade 3 or greater VLS. VLS will be dichotomized into absent or mild (grade 0-2) versus moderate to severe (3-5). Changes in FeNa from baseline to day 8, 10 and 12 will be calculated as percent change at each time point. Associations will be tested for in a logistic regression model using presence of moderate or severe VLS as outcome as well as in a linear regression model using the grading of VLS as an ordinal variable. Both models will be adjusted for the use of diuretics and intravenous fluids.
Maximum Plasma Concentration [Cmaxof CD19 and CD22 immunotxins will be measured | Pre-infusion; 4, 8, 12, 24 & 48 hours after start of the first and third infusion (course 1); pre-infusion and 4 hours after the start of the first and third infusions (subsequent courses)
  Maximum concentration (Cmax), t 1/2 (half-life), area under curve (AUC), and volume of distribution (Vd) will be determined. Serum concentrations of the immunotoxins will be measured and plotted against time. The association of the peak concentration (Cmax) with toxicities will be evaluated by using descriptive statistics and graphical methods.
Presence and percentage of bone marrow cells with a CD34+/CD38-/low/CD19+ phenotype | Up to day 42
  The presence of the postulated leukemic stem cells (LSC) with the CD34+/CD38-/low/CD19+ phenotype will be determined at baseline and after each cycle. A chi-square test or the non-parametric Fisher's exact test will be used to test for an association between the presence of the postulated LSC at baseline and/or after the first treatment cycle and response as the outcome. The analysis will be exploratory.
Presence of HAMA/HARA | Up to day 28 of course 1
  Tabulated or plotted by dose. HARA will only be determined after the first administration of Combotox (prior to course 2 and subsequent courses), whereas only HAMA will be determined prior to the first cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Verma, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Barta SK, Zou Y, Schindler J, Shenoy N, Bhagat TD, Steidl U, Verma A. Synergy of sequential administration of a deglycosylated ricin A chain-containing combined anti-CD19 and anti-CD22 immunotoxin (Combotox) and cytarabine in a murine model of advanced acute lymphoblastic leukemia. Leuk Lymphoma. 2012 Oct;53(10):1999-2003. doi: 10.3109/10428194.2012.679267. Epub 2012 Apr 18. PMID 22448921